CLINICAL TRIAL: NCT02360228
Title: Targeting Auditory Hallucinations With Alternating Current Stimulation
Brief Title: STimulation to Improve Auditory haLLucinations
Acronym: STILL 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14-3285; 1R21MH105574-01 (NIH)
Record Dates: First submitted 2015-02-02; First posted 2015-02-10 (Estimated); Results first posted 2018-04-27 (Actual); Last update posted 2018-04-27 (Actual); Status verified 2016-03

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: tACS; tDCS; sham; auditory hallucinations; Schizophrenia; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Hallucinations | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- tACS (alpha) (Experimental): 20 participants: 10Hz tACS with a peak-to-peak amplitude of 2mA for 20 minutes twice daily
  Interventions: Device: tACS (alpha)
- tDCS (Experimental): 20 participants: 2mA stimulation for 20 minutes twice daily
  Interventions: Device: tDCS
- Sham stimulation (Sham Comparator): 20 participants: Will include 10 seconds of ramp in to 1 minutes of 10 Hz tACS with a ramp out of 10 seconds for a total of 80 seconds of stimulation twice daily.
  Interventions: Device: tACS (alpha)

INTERVENTIONS:
Device: tACS (alpha)
  Arms: Sham stimulation; tACS (alpha)
Device: tDCS
  Arms: tDCS

SUMMARY:
Investigating the effects of non-invasive transcranial current stimulation as a treatment for auditory hallucinations in patients with schizophrenia.

DETAILED DESCRIPTION:
The investigator's primary objective is to conduct a pilot clinical trial to establish the feasibility and to collect first effectiveness data for the use of transcranial alternating current stimulation (tACS) to re-normalize pathological alpha oscillations in dorso-lateral prefrontal cortex (dl-PFC) of patients with schizophrenia or schizoaffective disorder by comparing Auditory Hallucination Rating Scale (AHRS) scores immediately before the first stimulation session and immediately after the last stimulation session. As a secondary objective the investigators will assess the differential clinical effects of sham, 10 Hz and 2 mA transcranial direct current stimulation (tDCS) on electroencephalogram (EEG) measures of alpha oscillations.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of schizophrenia, any subtype, or schizoaffective disorder, with refractory auditory hallucinations. Duration of illness >1 year
* 18-70 years old
* Clinically stable for at least 12 weeks, i.e. not requiring hospitalization or a change in level of care
* On current antipsychotic doses for at least 4 weeks
* Stable auditory hallucinations as demonstrated by having less than or equal to 20% change in AHRS scores across a 2 week interval during the screening period.
* Capacity to understand all relevant risks and potential benefits of the study and to provide written informed consent, OR has a legal guardian who can provide informed consent on the patient's behalf with the patient providing written assent to participate.

Exclusion Criteria:

* DSM-IV diagnosis of alcohol of substance abuse (other than nicotine) within the last month or a DSM-IV diagnosis of alcohol or substance dependence (other than nicotine) within the last 6 months
* Medical or neurological illness (unstable cardiac disease, AIDS, malignancy, liver or renal impairment) or treatment for a medical disorder that could interfere with study participation
* History of traumatic brain injury that required subsequent cognitive rehabilitation, or caused cognitive sequelae
* Prior brain surgery
* Any brain devices/implants, including cochlear implants and aneurysm clips
* Co-morbid neurological condition (e.g. seizure disorder, brain tumor)
* Non English speakers
* Female participants who are pregnant, nursing, or unwilling to use an adequate method of contraception during study participation for those of childbearing potential
* Positive urine test for cannabis, cocaine, amphetamine, barbiturates, benzodiazepines, opiates

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-05; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Flavio Frohlich, PhD, Principal Investigator — University of North Carolina at Chapel Hill - Department of Psychiatry
Locations (1):
- UNC Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- [Background] Brunelin J, Mondino M, Gassab L, Haesebaert F, Gaha L, Suaud-Chagny MF, Saoud M, Mechri A, Poulet E. Examining transcranial direct-current stimulation (tDCS) as a treatment for hallucinations in schizophrenia. Am J Psychiatry. 2012 Jul;169(7):719-24. doi: 10.1176/appi.ajp.2012.11071091. PMID 22581236

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited through medical providers or ads. Providers knew study criteria and discussed the study with patients during regular appointments. Interested participants contacted the study team, or were contacted by study team. Participants recruited from STEP clinic, Chapel Hill and Raleigh, and local clinics. Recruitment 4/15 to 12/16.
Pre-assignment Details: Participants randomly assigned to 1 of 3 arms, tDCS, tACS, or active sham. tDCS, tACS current delivered during awake, resting state for 20 minutes twice daily on 5 consecutive days. Sham stimulation was delivered for equal period of time and number of sessions. 33 participants signed consent, 7 screen fails, 1 withdrew.
Groups:
- tACS (Alpha): 10Hz transcranial alternating current stimulation (tACS) at the alpha frequency with a peak-to-peak amplitude of 2mA for 20 minutes twice daily
  tACS (alpha)
- tDCS: 2mA transcranial direct current stimulation (tDCS) for 20 minutes twice daily
- Sham Stimulation: Will include 10 seconds of ramp in to 1 minutes of 10 Hz tACS with a ramp out of 10 seconds for a total of 80 seconds of stimulation twice daily.
Period: Overall Study
Arm/Group | tACS (Alpha) | tDCS | Sham Stimulation
Started | 9 | 8 | 8
Completed | 8 | 7 | 7
Not Completed | 1 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Self-discontinued medication | 0 | 1 | 0
Not completed — Unstable symptoms during screening | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- tACS (Alpha): 10Hz tACS with a peak-to-peak amplitude of 2mA for 20 minutes twice daily
  tACS (alpha)
- tDCS: 2mA stimulation for 20 minutes twice daily
  tDCS
- Sham Stimulation: Will include 10 seconds of ramp in to 1 minutes of 10 Hz tACS with a ramp out of 10 seconds for a total of 80 seconds of stimulation twice daily.
  tACS (alpha)
- Total: Total of all reporting groups
Arm/Group | tACS (Alpha) | tDCS | Sham Stimulation | Total
Number analyzed (Participants) | 8 | 7 | 7 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (9.72) | 29.75 (10.97) | 38.86 (10.01) | 38.86 (12.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 3 | 7
  Male | 7 | 4 | 4 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 7 | 5 | 20
  Unknown or Not Reported | 0 | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 6 | 3 | 2 | 11
  White | 2 | 4 | 4 | 10
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 7 | 7 | 22
Auditory Hallucination Rating Scale [Mean (Standard Deviation); unit: units on a scale] — The Auditory Hallucination Rating Scale (AHRS) measures the severity of auditory hallucinations in the past week. The scale assesses frequency, duration, location, loudness, belief of origin of voices, negative content, distress, disruption to life, and control over voices. All items are measured on a scale of 0 to 4, with a total possible score of 44. Higher scores indicate higher severity of auditory hallucinations.
  units on a scale | 25.88 (3.80) | 23.00 (6.90) | 24.71 (5.91) | 24.59 (5.47)
Positive and Negative Syndrome Scale [Mean (Standard Deviation); unit: units on a scale] — The Positive and Negative Syndrome Scale (PANSS) is a clinical measure assessing the positive, negative, and general symptoms of psychosis. There are 30 items (7 positive, 7 negative, and 16 general). The score for each item ranges from 1 (absent) to 7 (extreme) and the PANSS total score ranges from 30 to 210, with higher scores indicating more severe symptoms.
  units on a scale | 52.75 (7.74) | 58.86 (14.66) | 57.00 (11.60) | 56.05 (11.27)
Brief Assessment of Cognition in Schizophrenia [Mean (Standard Deviation); unit: units on a scale] — The Brief Assessment of Cognition in Schizophrenia (BACS) is a battery of cognitive assessments assessing verbal memory and learning, working memory, motor function, verbal fluency, speed of processing, and executive function. Higher scores indicate better cognitive performance.
  Verbal Memory: Score out of 75
  Digit Sequencing: Score out of 28
  Token Motor: Score out of 100
  Fluency: No score limit
  Symbol Coding: Score out of 110
  Tower of London: Score out of 22
  Reported score is the mean of these 6 subtests. Healthy controls (Keefe et al., 2006) scored 45.6 as a comparison.
  units on a scale | 31.21 (5.68) | 38.26 (9.01) | 38.93 (7.17) | 35.91 (7.87)

OUTCOME MEASURES:

1. Primary Outcome: Proportional Change From Baseline in Auditory Hallucination Rating Scale (AHRS) Score
Description: The Auditory Hallucination Rating Scale (AHRS) measures the severity of auditory hallucinations in the past week. The scale assesses frequency, duration, location, loudness, belief of origin of voices, negative content, distress, disruption to life, and control over voices. All items are measured on a scale of 0 to 4, with a total possible score of 44. Higher scores indicate higher severity of auditory hallucinations. The investigators will compare the AHRS scores from immediately before the first stimulation and immediately after the last stimulation session as the investigator's primary outcomes measure.
Time Frame: Baseline, five days post baseline, 2 weeks post baseline, 5 weeks post baseline
Population: Per protocol; All eligible participants who completed every session of the study from the initial session through the one month follow-up that followed study protocol.
Measure: Mean (Standard Deviation); unit: proportion to baseline
Arm/Group | tACS (Alpha) | tDCS | Sham Stimulation
Number analyzed (Participants) | 8 | 7 | 7
proportion to baseline
  5 days from baseline | 0.85 (0.13) | 0.94 (0.36) | 0.91 (0.08)
  2 weeks from baseline | 0.84 (0.19) | 0.94 (0.20) | 0.92 (0.11)
  5 weeks from baseline | 0.85 (0.16) | 1.01 (0.14) | 0.85 (0.09)
Statistical Analysis 1: Comparison: tACS (Alpha) vs tDCS vs Sham Stimulation; The null hypothesis was that there is no difference between the changes in the AHRS score from baseline to 5 days between the groups.H0: μ1=μ2=μ3 μ1: mean(difference 5 days-baseline) for tACS group (n=8) μ2: mean(difference 5 days-baseline) for tDCS group (n=7) μ3: mean(difference 5 days-baseline) for sham group (n=7); Test type: Other; p = 0.47, ANOVA; Difference from day 5 to baseline was compared between the tACS, tDCS, and sham groups using a one way ANOVA. Degrees of freedom: df=19

2. Secondary Outcome: Change in Alpha Oscillations Measured With Electroencephalogram (EEG) Resting State From Baseline
Description: The investigators will compare alpha oscillation power from resting state EEG recordings on the first and last day of stimulation. The investigators will also collect EEG recordings data at the one week and one month follow up visits. The investigators will use each of the four EEG recordings as data to analyze alpha frequency activity as a pilot study for derivation of EEG biomarkers.
Time Frame: Baseline, five days post baseline
Population: Per protocol; All eligible participants who completed every session of the study from the initial session through the one month follow-up that followed the study protocol.
Measure: Mean (Standard Deviation); unit: decibel (dB)
Arm/Group | tACS (Alpha) | tDCS | Sham Stimulation
Number analyzed (Participants) | 8 | 7 | 7
decibel (dB) | 1.5 (0.2) | 0.3 (0.1) | 0.4 (0.2)

3. Secondary Outcome: Change in Positive and Negative Syndrome Scale (PANSS) Scores
Description: The investigators will compare the PANSS total scores immediately before first stimulation session and immediately after last stimulation session as secondary outcome measures. Scores range from 30 to 210, with higher scores indicating more severe symptomology.
Time Frame: baseline, five days post baseline, five weeks post baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | tACS (Alpha) | tDCS | Sham Stimulation
Number analyzed (Participants) | 8 | 7 | 7
scores on a scale
  5 days from baseline | 51.25 (8.19) | 54.71 (11.84) | 55.29 (10.86)
  5 weeks from baseline | 51.13 (9.95) | 52.86 (7.47) | 51.57 (12.20)
Statistical Analysis 1: Comparison: tACS (Alpha) vs tDCS vs Sham Stimulation; The null hypothesis was that there is no difference between the changes in the PANSS score from day 5 to baseline. H0: μ1=μ2=μ3 μ1: mean(difference 5 days-baseline) for tACS group (n=8) μ2: mean(difference 5 days-baseline) for tDCS group (n=7) μ3: mean(difference 5 days-baseline) for sham group (n=7); Test type: Other; p = 0.37, ANOVA; Difference from day 5 to baseline was compared between the tACS, tDCS, and sham using a one way ANOVA. Degrees of freedom: df=19

4. Secondary Outcome: Change in Brief Assessment of Cognition in Schizophrenia (BACS) Score
Description: The Brief Assessment of Cognition in Schizophrenia (BACS) is a battery of cognitive assessments assessing verbal memory and learning, working memory, motor function, verbal fluency, speed of processing, and executive function. Higher scores indicate better cognitive performance. The investigators will compare the BACS total scores immediately before first stimulation session and immediately after last stimulation session as secondary outcome measures.
  Verbal Memory: Score out of 75
  Digit Sequencing: Score out of 28
  Token Motor: Score out of 100
  Fluency: No score limit
  Symbol Coding: Score out of 110
  Tower of London: Score out of 22
  Reported score is the mean of these 6 subtests. Healthy controls (Keefe et al., 2006) scored 45.6 as a comparison.
Time Frame: baseline, five days post baseline, five weeks post baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | tACS (Alpha) | tDCS | Sham Stimulation
Number analyzed (Participants) | 8 | 7 | 7
scores on a scale
  5 days from baseline | 31.58 (5.77) | 42.05 (10.82) | 41.50 (10.52)
  5 weeks from baseline | 29.81 (5.50) | 39.71 (9.39) | 40.83 (9.71)
Statistical Analysis 1: Comparison: tACS (Alpha) vs tDCS vs Sham Stimulation; The null hypothesis was that there is no difference between the changes in the BACS score from baseline to 5 days between the groups: H0: μ1=μ2=μ3 μ1: mean(difference 5 days-baseline) for tACS group (n=8) μ2: mean(difference 5 days-baseline) for tDCS group (n=7) μ3: mean(difference 5 days-baseline) for sham group (n=7); Test type: Other; p = 0.11, ANOVA; [statistical method as in outcome 1, analysis 1]

5. Other Pre Specified Outcome: Change in Electroencephalogram (EEG) Auditory Tasks: Oddball Task From Baseline
Description: The investigators will compare auditory responses during auditory tasks EEG recordings on the first and last day of stimulation. The investigators will also collect EEG recordings data at the one week and one month follow up visits. The investigators will use each of the four EEG recordings as data to analyze alpha frequency activity as a pilot study for derivation of EEG biomarkers and look for increase in auditory responses.
  Auditory oddball paradigm is an experimental design that has standard (low-pitch) and deviant (high-pitch) stimuli. Differences in ERP from these two stimuli can measure functions of sensory processing. Patients with schizophrenia often exhibit abnormal responses to the stimuli thus its discrepancy compared to healthy human participants can be a hallmark of symptoms in schizophrenia.
Time Frame: baseline, five days post baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: micro volts
Arm/Group | tACS (Alpha) | tDCS | Sham Stimulation
Number analyzed (Participants) | 8 | 7 | 7
micro volts
  standard tones | 0.6 (0.1) | 0.4 (0.1) | 0.5 (0.1)
  deviant tones | 0.3 (0.05) | 0.4 (0.1) | 0.3 (0.1)

6. Other Pre Specified Outcome: Change in Electroencephalogram (EEG) Auditory Tasks: Click Train Task From Baseline
Description: The investigators will compare auditory responses during auditory tasks EEG recordings on the first and last day of stimulation. The investigators will also collect this data at the one week and one month follow up visits.
  Auditory steady-state response (ASSR) from EEG data elicited by auditory click trains is considered as a hallmark of network dysfunction in schizophrenia. To obtain ASSR, auditory tones at a specific frequency (e.g., 40Hz) are presented for multiple trials and EEG data is analyzed to extract brain responses to the stimuli.
  One common way to extract the brain responses from this task is phase coherence between trials. When external stimuli (click trains) occur, brain signals are synchronized to these stimuli and its coherence should be the highest at the stimulation frequency. Phase information for calculating the coherence can be obtained by time-frequency analysis. Averaged coherence across the multiple trials can represent the inter-trial phase coherence.
Time Frame: baseline, five days post baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: inter-trial phase coherence
Arm/Group | tACS (Alpha) | tDCS | Sham Stimulation
Number analyzed (Participants) | 8 | 7 | 7
inter-trial phase coherence
  topographical activity | 5 (0.1) | 0.5 (0.1) | 0.5 (0.1)
  time-frequency activity | 1 (0.01) | 0.05 (0.01) | 0.04 (0.01)

7. Secondary Outcome: Change in Peak Frequency of Functional Connectivity From Baseline Measured With Electroencephalogram (EEG) Resting State
Description: The investigators will compare peak frequency of functional connectivity from resting state EEG recordings on the first and last day of stimulation. The investigators will also collect EEG recordings data at the one week and one month follow up visits. The investigators will use each of the four EEG recordings as data to analyze the change in peak frequency of functional connectivity as a pilot study for derivation of EEG biomarkers.
Time Frame: Baseline, five days post baseline
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Hertz (Hz)
Arm/Group | tACS (Alpha) | tDCS | Sham Stimulation
Number analyzed (Participants) | 8 | 7 | 7
Hertz (Hz) | 10 (0) | 8 (0.5) | 11 (0.5)

ADVERSE EVENTS:
Time Frame: Adverse events data collected from the beginning of the study (6/2015) through the completion of the study (2/2017) for a total of 20 months.
Arm/Group | tACS (Alpha) | tDCS | Sham Stimulation
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 0/8 | 0/7 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-04-29): https://cdn.clinicaltrials.gov/large-docs/28/NCT02360228/Prot_SAP_000.pdf